CLINICAL TRIAL: NCT02791594
Title: Imaging the Flare Response With FDG PET/CT in Patients With Advanced Metastatic Melanoma on Pembrolizumab.
Brief Title: Imaging FDG Flare in Melanoma
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: UPCC 02616
Record Dates: First submitted 2016-06-01; First posted 2016-06-07 (Estimated); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pembrolizumab — Patients were treated with pembrolizumab according to standard of care.

SUMMARY:
Up to 35 adult patients with metastatic melanoma planning to start pembrolizumab will be enrolled in this study with a target enrollment of 30 evaluable subjects. Subjects will complete a baseline FDG PET/CT and an on-treatment FDG PET/CT after 1 week of pembrolizumab therapy. Subjects may also be a part of the Penn Melanoma Tissue Collection Program and then will be asked to have one additional tumor biopsy and one additional blood draw for the purposes of this imaging study. Changes in tumor FDG uptake between the baseline and early on-treatment FDG PET/CT scans will be correlated with blood and tissue results from the patient's medical records and from the data collected as part of the Penn Melanoma Tissue Collection Program and with outcomes including objective response, progression free survival, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures.
* The subject must be ≥ 18 years of age on day of signing informed consent.
* The subject must have biopsy proven or clinically documented advanced stage metastatic melanoma.
* The subject must have measurable disease (per RECIST 1.1) that is seen on CT, MRI, or FDG PET/CT.
* The subject must be recommended to start pembrolizumab.

Exclusion Criteria:

* Females who are pregnant or breast-feeding at the time of screening will not be eligible for this study. Female participants of child-bearing potential will have a urine pregnancy test at the time of the screening visit.
* Subject is not able to tolerate imaging procedures in the opinion of the investigator or treating physician.
* Subject has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Subject has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent as assessed by medical record review and/or self-reported.
* Subject has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) as determined by medical record review.
* Subject has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Subject has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected) as determined by medical record review.
* Subject has known active central nervous system metastases and/or carcinomatous meningitis.

Note: Subjects with previously treated brain metastases will be eligible to participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to receiving pembrolizumab and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Melanoma
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2016-06; Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Farwell, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Early FDG PET/CT Imaging Group: Patients with advanced melanoma (Stage 3B - Stage 4) scheduled to be treated with pembrolizumab had a baseline 18F-fluorodeoxyglucose (FDG) PET/CT scan (PET0) at a median of 9 days (range, 0 - 24 days) prior to initiation of pembrolizumab, and a follow-up FDG PET/CT scan (PET1) at a median of 7 days (range, 3 - 21 days) after the first dose of pembrolizumab.
Period: Overall Study
Arm/Group | Early FDG PET/CT Imaging Group
Started | 21
Completed | 19
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Early FDG PET/CT Imaging Group
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 19
Cancer Stage [Count of Participants; unit: Participants] — Stage 3 melanoma has spread to regional lymph nodes or has developed in-transit deposits of disease, but there is no evidence of distant metastasis; stage 3C melanoma is more advanced compared to Stage 3B. Stage 4 melanoma has traveled beyond the original tumor site and beyond the regional lymph nodes to more distant sites in the body.
  Participants
    Stage 3B | 2
    Stage 3C | 4
    Stage 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Objective Response by RECIST Version 1.1
Description: Objective response is defined as the proportion of patients with a complete response or partial response by RECIST version 1.1. A complete response is defined as the disappearance of all tumor lesions, and a decrease in size of all pathological lymph nodes to <10 mm along the short axis. A partial response is at least a 30% decrease in the sum of diameters of target tumor lesions, taking as reference the baseline sum diameters.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Early FDG PET/CT Imaging Group
Number analyzed (Participants) | 19
Participants
  Responders (complete response + partial response) | 11
  Non-responders (progressive disease or pathologic non-response) | 8

2. Primary Outcome: Number of Participants With Change in Tumor FDG Uptake Between Baseline FDG PET/CT and Early On-Treatment FDG PET/CT Obtained 1 Week After Initiation of Pembrolizumab
Description: FDG PET scans were evaluated for changes in maximum standardized uptake value (SUVmax) for up to 5 RECIST-measurable lesions (2 per organ) for each patient. The percentage change in SUVmax was defined as (sum of PET1 SUVmax - sum of PET0 SUVmax)/(sum of PET0 SUVmax) x 100, where PET0 was the baseline FDG PET/CT and PET1 was the on-treatment FDG PET/CT acquired at ~1 week after starting pembrolizumab. A metabolic flare (MF) was defined as >70% increase in tumor SUVmax between baseline and follow-up scans, and a metabolic response (MR) was defined as a >30% decrease in tumor SUVmax. If the change in tumor SUVmax was neither MF or MR it was classified as stable metabolism (SM).
Time Frame: Baseline and 1 week after initiation of pembrolizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Early FDG PET/CT Imaging Group
Number analyzed (Participants) | 19
Participants
  Metabolic Flare or Metabolic Response | 6
  Stable Metabolism | 13

3. Secondary Outcome: Progression-Free Survival
Description: Progression-Free Survival is defined as time from the PET1 scan (acquired 1 week after starting pembrolizumab) to progression, according to RECIST 1.1, or death from any cause, whichever occurs first. Patients who neither progress nor die during the study will be censored at the date of last disease assessment without progression.
Time Frame: 4 years
Population: The overall number of participants analyzed is 19, but the progression-free survival was calculated for each cohort: MF-MR cohort (6 participants) and SM cohort (13 participants).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Early FDG PET/CT Imaging Group
Number analyzed (Participants) | 19
months
  MF-MR cohort: number analyzed (Participants) | 6
  MF-MR cohort | NA [NA to NA] — Median PFS was not reached in this cohort (but was >38 months) because there were an insufficient number of participants with events.
  SM cohort: number analyzed (Participants) | 13
  SM cohort | 2.8 [0.3 to 5.2]

4. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) was defined as time from the PET1 scan (6-10 days after start of immunotherapy) to death from any cause, with patient censoring at date last known alive.
Time Frame: 4 years
Population: The overall number of participants analyzed is 19, but the overall survival was calculated for each cohort: MF-MR cohort (6 participants) and SM cohort (13 participants).
Measure: Number; unit: percentage of patients that died
Arm/Group | Early FDG PET/CT Imaging Group
Number analyzed (Participants) | 19
percentage of patients that died
  MF-MR cohort: number analyzed (Participants) | 6
  MF-MR cohort | 17
  SM cohort: number analyzed (Participants) | 13
  SM cohort | 38

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored/assessed for up to 4 years. Adverse events were monitored/assessed for the period of time from the injection of FDG to the completion of the imaging exam (for 2 hours).
Description: Adverse events related to the standard of care clinical treatment (pembrolizumab) were not collected or reported as part of this study.
Arm/Group | Early FDG PET/CT Imaging Group
All-Cause Mortality (participants affected / at risk) | 6/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT02791594/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/94/NCT02791594/ICF_001.pdf